CLINICAL TRIAL: NCT01082120
Title: Open, Randomized, Phase I Study in Subjects With Type 2 Diabetes Mellitus Treated With Metformin to Evaluate the Effect of AZD1656 on the Pharmacokinetics of Pioglitazone and Vice Versa
Brief Title: Investigate the Effect of AZD1656 on the Pharmacokinetics of Pioglitazone and Vice Versa in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00028
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Pioglitazone
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD1656 day 1-5, AZD1656 + Pioglitazone day 6-10, Pioglitazone day 11-15
  Interventions: Drug: AZD1656; Drug: Pioglitazone
- 2 (Experimental): Pioglitazone day 1-5, AZD1656 + Pioglitazone day 6-10, AZD1656 day 11-15
  Interventions: Drug: AZD1656; Drug: Pioglitazone

INTERVENTIONS:
Drug: AZD1656 — Tablets orally, twice daily for 10 days
Drug: Pioglitazone — Tablet oral single dose for 10 days

SUMMARY:
The purpose of this study is to determine whether administration of AZD1656 will affect the pharmacokinetics of Pioglitazone and vice versa in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Type 2 Diabetes Mellitus for at least 1 year and treated with metformin alone or metformin and one other oral anti-diabetic drug
* Body mass index between ≥19 and ≤42 kg/m2.

Exclusion Criteria:

* Impaired renal function
* Clinically significant illness or clinically relevant trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of AZD1656 on the steady state pharmacokinetics of Pioglitazone and vice versa by assessment of AUC (0-24) and Cmax. | Serial blood samples on Days 5, 10 and 15 to assess pharmacokinetics of Pioglitazon, the metabolite hydroxyl-Pioglitazone, AZD1656 and its metabolite as appropriate.

SECONDARY OUTCOMES:
To evaluate the effect of AZD1656 on the steady state pharmacokinetics of Pioglitazone and vice versa by assessment of tmax, t1/2 and CL/F. | Serial blood samples on Days 5, 10 and 15 to assess pharmacokinetics of Pioglitazon, the metabolite hydroxyl-Pioglitazone, AZD1656 and its metabolite as appropriate.
To evaluate the pharmacokinetics of the AZD1656 and its metabolite, when AZD1656 is administered with and without pioglitazone, by assessment of AUC(0 24), Cmax and tmax. | Serial blood samples on Days 5, 10 and 15 to assess pharmacokinetics of Pioglitazon, the metabolite hydroxyl-Pioglitazone, AZD1656 and its metabolite as appropriate.
To evaluate the pharmacokinetics of the Pioglitazone metabolite hydroxyl pioglitazone, when pioglitazone is administered with and without AZD1656, by assessment of AUC(0-24), Cmax and tmax. | Serial blood samples on Days 5, 10 and 15 to assess pharmacokinetics of Pioglitazon, the metabolite hydroxyl-Pioglitazone, AZD1656 and its metabolite as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Stanko Skrtic, Study Director — AstraZeneca; Elaine Watkins, DO, Principal Investigator — Profil Institute for Clinical Research, Inc.; Mirjana Kujacic, Study Chair — AstraZeneca
Locations (1):
- Research Site, Chula Vista, California, United States